CLINICAL TRIAL: NCT00623298
Title: Narrative Exposure Therapy Versus Group Interpersonal Psychotherapy -A Controlled Clinical Trial With Orphaned Survivors of the Rwandan Genocide
Brief Title: Narrative Exposure Therapy Versus Group Interpersonal Psychotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: vivo (Unknown)
Responsible Party: Dr. Susanne Schaal, University of Konstanz, vivo
Allocation: Non-Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: Fogr SOSS
Record Dates: First submitted 2008-02-14; First posted 2008-02-26 (Estimated); Last update posted 2008-02-26 (Estimated); Status verified 2008-02

CONDITIONS: Posttraumatic Stress Disorder; Depression; Narrative Exposure Therapy; Interpersonal Psychotherapy
Keywords: Posttraumatic stress disorder; depression; Narrative Exposure Therapy; Interpersonal Psychotherapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression | interventions — BaseLine dental cement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): NET
  Interventions: Behavioral: Narrative Exposure Therapy
- 3 (No Intervention): 6-months baseline
  Interventions: Other: 6 months-baseline
- 2 (Experimental): group IPT
  Interventions: Behavioral: group IPT

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy
  Arms: 1
Behavioral: group IPT
  Arms: 2
Other: 6 months-baseline
  Arms: 3

SUMMARY:
The present study is a pragmatic trial that investigates the efficacy and usefulness of two treatment modules in a sample of Rwandan genocide orphans: Narrative Exposure Therapy (NET) versus group-Interpersonal Psychotherapy (IPT). We used a half year baseline to measure the treatment-induced changes. We hypothesized that there would be a greater reduction in posttraumatic stress symptoms in the NET- than in the IPT-group and that IPT would be superior to NET in the reduction of depression symptoms.

DETAILED DESCRIPTION:
The 1994 genocide of Rwanda has left countless children orphaned. 26 Rwandan orphans who fulfilled DSM-IV diagnosis of PTSD were offered participation in a controlled treatment trial. A group adaptation of Interpersonal Psychotherapy (IPT, n = 14) was compared to Narrative Exposure Therapy (NET, n = 12). Main outcome measures were symptoms of PTSD and depression assessed pre-treatment, 3 months after therapy (post-test) and 6 months after therapy (follow-up) using the CAPS, MINI and Hamilton Rating Scale. At post-test, participants in both treatment conditions showed reductions in posttraumatic stress symptoms and depression symptoms. At 6-month follow-up, NET proved to be more effective in the treatment of PTSD. Only 25% (n = 3) of NET-participants but 71% (n = 10) of the IPT-participants still fulfilled PTSD criteria at follow-up. Although there was a significant reduction in depression symptoms in both treatment groups from pre-test to follow-up, NET again proved to be more effective. This treatment-trial demonstrates that NET and group-IPT are suitable treatment modules even when most severe traumatic stress and difficult living conditions have led to chronic mental suffering.

ELIGIBILITY:
Inclusion Criteria:

* Rwandan orphans who have experienced the genocide, who lost at least one parent during the genocide and who were no older than 18 years during the genocide

Exclusion Criteria:

* Mental retardation
* Psychotic symptoms or current drug or alcohol

Ages: 13 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2005-01; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Symptoms of posttraumatic stress disorder, symptoms of depression